CLINICAL TRIAL: NCT04170140
Title: A Cross-sectional Survey to Evaluate Prescribers' Knowledge and Understanding of Safety Messages Following Dengvaxia® Product Information Update
Brief Title: Study on Prescribers' Knowledge and Understanding of Safety Messages Following Dengvaxia® Product Information Update
Acronym: DNG00042
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DNG00042; U1111-1233-9599 (Other: UTN)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-04

CONDITIONS: Dengue Virus Infection
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prescribers of Dengvaxia: Healthcare professionals who are current or past prescribers of Dengvaxia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Questionnaire

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of additional risk minimization measures material by assessing the knowledge and understanding of healthcare professionals regarding the key safety messages provided in the material.

The secondary objective of the study is to evaluate if healthcare professionals know Dengvaxia product information, namely, age indication and contraindications.

DETAILED DESCRIPTION:
The study is a cross-sectional Survey. Study data are collected through a questionnaire.

ELIGIBILITY:
Inclusion criteria:

- Healthcare professionals who are current or past prescribers of Dengvaxia

Exclusion criteria:

* Healthcare professionals who have never prescribed Dengvaxia
* Healthcare professionals who may have a conflict of interest with the survey (i.e. Healthcare professionals employed by regulatory bodies, pharmaceutical industries)
* Healthcare professionales who have participated in testing the questionnaire for comprehensibility, consistency and the appropriateness of medical terms

The above information is not intended to contain all considerations relevant to participation in the survey.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals who are current or past prescribers of Dengvaxia
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Healthcare professionals' knowledge and understanding of key safety messages provided in risk minimization measures materials | Day 0
  Knowledge and understanding of key safety messages are assessed through a questionnaire

SECONDARY OUTCOMES:
Healthcare professionals' knowledge of Dengvaxia product information | Day 0
  Knowledge of Dengvaxia product information (age indication and contraindications) is assessed through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Real World Evidence Solutions IQVIA, La Defense, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Almas MF, Toussi M, Valero E, Moureau A, Marcelon L. A cross-sectional survey to evaluate prescribers' knowledge and understanding of safety messages following Dengvaxia(R) product information update. Pharmacoepidemiol Drug Saf. 2022 Jul;31(7):758-768. doi: 10.1002/pds.5447. Epub 2022 May 13. PMID 35505623